CLINICAL TRIAL: NCT04464486
Title: Remote COVID-19 Symptom Tracking and Improved Cancer Symptom Control for Cancer Patients at Home During the Pandemic
Brief Title: Remote COVID-19 Symptom Tracking for Cancer Patients at Home During the Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kathleen Mooney, Distinguished Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00131892
Record Dates: First submitted 2020-06-26; First posted 2020-07-09 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 Symptom Augmented SCH Intervention (Experimental): The SCH intervention group will report COVID-19 and cancer-related symptom presence and severity daily into the automated SCH system. Participants receive automated self-management support messages for symptoms reported and a Nurse Practitioner monitors and responds to alerts for COVID-19 symptoms and poorly controlled or worsening cancer symptoms. Participants in this group complete baseline and monthly measures.
  Interventions: Other: SCH Intervention
- Enhanced Usual Care (No Intervention): Participants in the control group are given information by research staff reviewing COVID-19 symptoms, home precautions, and instructions on what to do to address concerns that arise. Participants in this group complete baseline and monthly measures.

INTERVENTIONS:
Other: SCH Intervention — In addition to receiving usual care from their oncologist and staff, the SCH intervention group will report COVID-19 and cancer-related symptom presence and severity daily into the automated SCH system. Participants in the intervention receive automated self-management support messages for symptoms reported. In addition, COVID-19 symptoms and poorly controlled or worsening cancer symptoms will generate alerts. Based on preset thresholds, alerts automatically generate immediately from the patient's daily call data. The study nurse practitioners (NPs) monitor alerts. The NPs provide follow-up care using the guideline based SCH symptom clinical decision support system. The NPs log into the SCH Alert and Call Data website which displays all of the patients who have called that day and met an alert threshold. The NP calls the patient, delivers symptom management care by phone, and documents care in the patients' electronic health records.
  Other Names: Symptom Care at Home Intervention
  Arms: COVID-19 Symptom Augmented SCH Intervention

SUMMARY:
This project will evaluate the benefit of an automated home symptom monitoring system, Symptom Care at Home, to track COVID-19 symptoms, provide instructions to reduce COVID-19 exposure, and reduce cancer symptom severity during the COVID-19 pandemic. The investigators will determine if Symptom Care at Home decreases the need for cancer patients to use emergency departments and hospitalization for cancer symptom care. The project addresses the urgent public health need for cancer patients to reduce their risk for COVID-19 exposure.

DETAILED DESCRIPTION:
In response to the COVID-19 pandemic, there is an opportunity to rapidly flex platforms for remote cancer symptom tracking and management to incorporate COVID-19 symptom monitoring and reinforce risk-reducing precautions. It is critical for cancer patients at home to monitor early indications of COVID-19 symptoms, to adhere to mitigation strategies, as well as to manage their cancer-related symptoms so that patients can decrease the need to utilize the emergency department or unplanned hospitalizations for symptom care, which is a common occurrence during cancer care. Remote monitoring adds a layer of home-based support which can benefit all cancer patients and is not restricted to geographic proximity to oncology providers or distance from a cancer center. The Symptom Care at Home (SCH) system, utilized for the Principal Investigator's currently funded R01CA206522 project to monitor and manage patient-reported (PRO) cancer symptoms, includes these necessary elements: remote PRO symptom monitoring, patient self-management information, and oncology provider (nurse practitioner) notification of symptoms exceeding pre-set thresholds. The overall purpose of this project is to describe the impacts of COVID-19 on cancer patients' well-being at home and evaluate, through a randomized clinical trial, if a systematic patient-reported outcomes (PRO) reporting process improves cancer care during a pandemic as compared to usual care. Specific Aims include: 1) describe patient-reported COVID-19 and cancer symptom trajectories over time, COVID-19 social distancing and hygiene practices, and COVID-19 related cancer treatment and daily living impacts on cancer patients receiving the SCH-COVID intervention and 2) compare the SCH-COVID intervention to enhanced usual care on health care utilization, COVID-19 diagnosis and outcomes, cancer treatment delays or changes, and patient-reported global health, anxiety, mood, and feelings of social isolation.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be patients who are receiving treatment for a cancer diagnosis at Huntsman Cancer Hospital.
* Must be able to speak, read, and understand English language.
* Must have a smartphone and be willing and able to download the SCH application and enter data into the application OR must be willing to make phone calls to report symptoms using the telephone interactive voice response (IVR) system.

Exclusion Criteria:

* Patients enrolled in another study protocol that prohibits participation in other trials.
* Patients under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2020-04-21 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Health Care Utilization Comparison | 5 months
  Retrospective chart review of health care utilization of both groups

SECONDARY OUTCOMES:
Patient Social Isolation | Monthly for 5 months
  Patient Reported Outcomes Measurement Information System- Short Form v2.0 Social Isolation- 6a. The PROMIS Social Isolation item bank assesses perceptions of being avoided, excluded, detached, disconnected from, or unknown by, others. The item bank does not use a time frame (e.g. over the past seven days) when assessing social isolation. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like Social Isolation, a T-score of 60 is one SD worse than average. By comparison, a Social Isolation Tscore of 40 is one SD better than average.
COVID-19 Symptoms, Social distancing and Hygiene Practices | Daily for 5 months
  Patient reported outcomes collected in automated SCH system daily of COVID-19 symptoms, social distancing and hygiene practices, and COVID-19 related cancer treatment impacts and daily living impacts on cancer patients receiving the SCH -COVID intervention. The investigators will describe patterns of cancer patients and their adherence to social distancing and hygiene practices over time.
Patient Global Health | Monthly 5 months
  Patient Reported Outcomes Measurement Information System Scale v1.2- Global Health Survey Short Form 10. High scores reflect better functioning. To find the total raw score for these scales with all questions answered, sum the values of the response to each question for a given respondent.
Patient Anxiety/Depression | Monthly 5 months
  Hospital Anxiety and Depression Scale (HADS) measurement of psychological distress in non-psychiatric patients.
Impact of Pandemic and Health Related Quality of Life | Baseline then 3 months and 5 months from baseline
  COVID-19: Impact of the Pandemic and Health Related Quality Of Life (HRQOL) in Cancer Patients and Survivors
Cancer symptom severity | Daily for 5 months.
  Patient reported outcomes collected in automated SCH system daily of cancer symptom severity on a scale of 0-10 with 0 being no pain and 10 being worst pain imaginable. Description of symptom severity over time will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Mooney, PhD, Principal Investigator — University of Utah College of Nursing
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Secondary data analysis and use by other investigators is welcomed once the proposed aims have been analyzed and published. PI Mooney will share de-identified data with other investigators for study by proposing aims/hypotheses and identifying the data elements required and receiving agreement from the research team. Data will be shared with investigators working under an institution with a Federal Wide Assurance (FWA). The research team agrees to share data in a manner that is fully consistent with the data sharing policies of NIH and the University of Utah as well as applicable laws and regulations.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After acceptance of the main findings publications in peer reviewed scientific journals.
Access Criteria: Data will be available to address research questions/hypothesis of the request. Once the Principal Investigator reviews the research question proposed, the data elements that can address the question will be shared.